CLINICAL TRIAL: NCT01128179
Title: A Proof of Concept, Phase 2a, Double-blind, Parallel Group, Randomised, Placebo-controlled Study to Assess the Effect of Lanthanum Carbonate on Intact FGF23 in Normo-phosphataemic Subjects With Stage 3 Chronic Kidney Disease
Brief Title: Effects of Lanthanum Carbonate on FGF-23 in Subjects With Stage 3 CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD405-703; 2009-016531-35 (EudraCT Number)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lanthanum carbonate (Experimental)
  Interventions: Drug: Lanthanum carbonate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanthanum carbonate — 1000 mg in chewable tablets administered three times a day (for a total of 3000 mg/day) for 12 weeks
  Other Names: Fosrenol/Foznol
  Arms: Lanthanum carbonate
Drug: Placebo — Matching placebo chewable tablets administered 3 times a day for 12 weeks
  Arms: Placebo

SUMMARY:
To assess the effects of 12 weeks of treatment with lanthanum carbonate compared with placebo on serum intact Fibroblast Growth Factor 23 (FGF23) levels.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the criteria listed below may be included in the study:

1. ≥18 years old.
2. Male, or non-pregnant, non-lactating females who agree to comply with any applicable contraceptive requirements of the protocol.
3. Been in the care of a physician for CKD for >2 months, and are not expected to begin dialysis for at least 6 months.
4. Screening serum c-terminal FGF23 > 50.0RU/mL.
5. Screening estimated glomerular filtration rate (eGFR) of 30-59mL/min/1.73m2 using the MDRD formula.
6. Normal serum phosphate (0.808-1.55mmol/L).
7. Endogenous 25-hydroxy Vitamin D levels >20ng/mL.
8. Adequate protein diet (includes 2-3 portions of protein-rich food per day).
9. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
10. Ability to provide written, signed, and dated (personally) informed consent to participate in the study.

Exclusion Criteria

1. Vitamin D supplementation required.
2. Compounds containing calcium, phosphate, aluminium or magnesium required.
3. Acute renal failure.
4. Rapidly progressing glomerulonephritis.
5. Vegetarian diet.
6. Known allergy to iodine.
7. Clinically significant uncontrolled concurrent illness, which, in the opinion of the Investigator, would impair subjects' ability to give informed consent or take part in or complete this clinical study.
8. Cirrhosis or other clinically significant liver disease (aspartate transaminase (AST) or alanine transaminase (ALT) >3 times the upper limit of normal or bilirubin >2 times the upper limit of normal).
9. Past (treated within the last 5 years) or present GI disorders including uncontrolled peptic ulcer, Crohn's disease (or other conditions where the integrity of the GI tract may be compromised), malignancy, or GI bleed within the last 6 months.
10. Life-threatening malignancy or current multiple myeloma.
11. Known to be Human Immunodeficiency Virus (HIV) positive.
12. History of poor compliance with diet or medication that in the Investigator's opinion may interfere with adherence to the protocol.
13. History of alcohol or other substance abuse within 6 months prior to screening.
14. Subjects must not have used another investigational medicinal product or taken part in a clinical trial within the last 30 days prior to enrolment.
15. Subjects who have previously been enrolled into this study and subsequently withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-12-06 (Actual); Primary Completion 2012-04-16 (Actual); Study Completion 2012-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Dr Pablo Urena Torres, Saint-Ouen, Paris, France

REFERENCES:
- [Result] Urena-Torres P, Prie D, Keddad K, Preston P, Wilde P, Wan H, Copley JB. Changes in fibroblast growth factor 23 levels in normophosphatemic patients with chronic kidney disease stage 3 treated with lanthanum carbonate: results of the PREFECT study, a phase 2a, double blind, randomized, placebo-controlled trial. BMC Nephrol. 2014 May 5;15:71. doi: 10.1186/1471-2369-15-71. PMID 24885942
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanthanum Carbonate: 1000 mg in chewable tablets (given as 2 x 500 mg tablets) administered three times a day (for a total of 3000 mg/day) for 12 weeks
Period: Overall Study
Arm/Group | Lanthanum Carbonate | Placebo
Started | 23 | 12
Completed | 21 | 12
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was defined as all randomized subjects who received at least 1 dose of investigational product. This population was used in all safety reporting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate | Placebo | Total
Number analyzed (Participants) | 23 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (13.9) | 69.4 (13.2) | 67.2 (13.6)
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 23 | 12 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 13 | 5 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  France | 23 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Natural Logarithm Transformed Serum Intact Fibroblast Growth Factor (FGF-23) Levels at Week 12 Last Observation Carried Forward (LOCF)
Description: FGF-23 plays an important role in mineral metabolism in chronic kidney disease patients. It is secreted by bone cells in response to hyperphosphatemia. It acts to decrease renal phosphate reabsorption. Administration of a phosphate-binder (i.e. lanthanum carbonate) was expected to produce a reduction in FGF-23 levels.
Time Frame: 12 Weeks
Population: Per-protocol (PP) set are subjects who received at least 1 dose of investigational product and who had primary data assessment available from Week 2 or later and who did not have pre-defined major protocol deviations that could have affected the primary variable.
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
pg/ml | 4.0089 (0.0709) | 4.1210 (0.0844)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; Assuming that the natural logarithm transformed serum intact FGF-23 is normally distributed with a mean of 3.5 and a standard deviation of 0.46, 33 subjects randomised 2:1 (lanthanum carbonate to placebo) will be sufficient to detect with 80% power at the 5% 2-sided significance level a decrease of 0.5 in the mean difference (placebo minus lanthanum carbonate) of the log-transformed data at Week 12; Test type: Superiority or Other; p = 0.3186, ANCOVA — The a priori significance level was 5%. There was no adjustment for multiple comparisons; Mean Difference (Final Values) = -0.1121, 95% CI 2-sided [-0.3389 to 0.1146]

2. Secondary Outcome: Change From Baseline in Serum Intact Parathyroid Hormone (iPTH) Values at Week 12 (LOCF)
Time Frame: 12 Weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
pg/ml | 1.67 (3.96) | -4.87 (4.72)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of serum iPTH at Week 12 (LOCF) in an analysis of covariance (ANCOVA) with treatment as a factor and the baseline iPTH as a covariate. The study was not powered for the analysis of this parameter; Test type: Superiority or Other; p = 0.2995, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = 6.54, 95% CI 2-sided [-6.15 to 19.23]

3. Secondary Outcome: Change From Baseline in 1,25-Dihydroxy Vitamin D Values at Week 12 (LOCF)
Time Frame: 12 weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
pg/ml | -1.75 (3.22) | -6.86 (3.85)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of 1,25-Dihydroxy Vitamin D at Week 12 (LOCF) when utilizing an analysis of covariance (ANCOVA) with treatment as a factor and the baseline 1,25-Dihydroxy Vitamin D as a covariate. The study was not powered for the analysis of this parameter; Test type: Superiority or Other; p = 0.3252, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [-5.36 to 15.57]

4. Secondary Outcome: Change From Baseline in Urinary Fractional Excretion of Phosphate Values at Week 12 (LOCF)
Time Frame: 12 weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: percentage of excretion of phosphate
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
percentage of excretion of phosphate | -5.9 (1.5) | -2.2 (1.9)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of Urinary Fractional Excretion of Phosphate at Week 12 (LOCF) when utilizing an analysis of covariance (ANCOVA) with treatment as a factor and the baseline Urinary Fractional Excretion of Phosphate as a covariate. The study was not powered for the analysis of this parameter; Test type: Superiority or Other; p = 0.1459, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-8.845 to 1.403]

5. Secondary Outcome: Change From Baseline in Serum Phosphate Values at Week 12 (LOCF)
Time Frame: 12 weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
mmol/L | 0.0053 (0.0371) | 0.0350 (0.0443)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of Serum Phosphate at Week 12 (LOCF) in an analysis of covariance (ANCOVA) with treatment as a factor and the baseline Serum Phosphate as a covariate. The study was not powered for the analysis of this parameter; Test type: Superiority or Other; p = 0.6134, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = -0.0297, 95% CI 2-sided [-0.1492 to 0.0897]

6. Secondary Outcome: Change From Baseline in Serum Total Calcium Values at Week 12 (LOCF)
Time Frame: 12 weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
mmol/L | 0.0242 (0.0323) | -0.0052 (0.0385)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of Serum Total Calcium at Week 12 (LOCF) in an analysis of covariance (ANCOVA) with treatment as a factor and the baseline Serum Total Calcium as a covariate. The study was not powered for the analysis of this parameter; Test type: Superiority or Other; p = 0.5636, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = 0.0294, 95% CI 2-sided [-0.0739 to 0.1328]

7. Secondary Outcome: Change From Baseline in Calcium-Phosphate Product Values at Week 12 (LOCF)
Time Frame: 12 weeks
Population: PP
Measure: Least Squares Mean (Standard Error); unit: mmol^2/L^2
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 12
mmol^2/L^2 | 0.0581 (0.0833) | 0.0710 (0.0993)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Placebo; The null hypothesis was that there would be no difference between the 2 treatment groups in the mean change from baseline of Calcium-Phosphate Product at Week 12 (LOCF) in an analysis of covariance (ANCOVA) with treatment as a factor and the baseline Calcium-Phosphate Product as a covariate; Test type: Superiority or Other; p = 0.9220, ANCOVA — The p-value was unadjusted and had no a priori significance level; Mean Difference (Final Values) = -0.0129, 95% CI 2-sided [-0.2811 to 0.2553]

ADVERSE EVENTS:
Arm/Group | Lanthanum Carbonate | Placebo
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/12
Other Adverse Events (participants affected / at risk) | 2/23 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanthanum Carbonate (N=23) | Placebo (N=12)
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanthanum Carbonate (N=23) | Placebo (N=12)
Constipation (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.